CLINICAL TRIAL: NCT04199728
Title: Use of a GLP-1R Agonist to Treat Opioid Use Disorder
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Scott C Bunce, PhD, Associate Professor of Psychiatry, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13559; 1UG3DA050325-01 (NIH)
Record Dates: First submitted 2019-12-12; First posted 2019-12-16 (Actual); Results first posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Opiate Substitution Treatment; Opioid-Related Disorders
Keywords: Opiate treatment; Opioid treatment; Glucagon-Like Peptide-1 Agonist; Opioid use disorder; Liraglutide
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Investigational group (Experimental): Participants randomized to liraglutide will be started at a low dose (0.6 mg once per day) which will be gradually increased until 1.8 mg/day is reached for the 3-dose intervention and 3 mg/day is reached for the 5-dose intervention. Liraglutide will be administered by injection pen.
  Interventions: Drug: Liraglutide Pen Injector
- Control group (Placebo Comparator): Participants in the control group will have placebo administered by injection pen following the same low dose titration to 3.0 mg once per day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Liraglutide Pen Injector — Liraglutide will be provided using an injection pen provided by the manufacturer
  Other Names: Saxenda
  Arms: Investigational group
Drug: Placebo — Placebo injection pen
  Arms: Control group

SUMMARY:
This research is being done to find out if liraglutide (brand name is Saxenda®) can safely and effectively reduce craving for opioids in patients with opioid use disorder, a primary factor contributing to early relapse.

DETAILED DESCRIPTION:
The rationale for the proposed research is to develop an acute intervention that can improve treatment outcomes in opioid use disorder (OUD) by reducing craving, a primary factor contributing to early relapse. Although liraglutide was approved for human use in 2010, there are no data testing the effectiveness in patients with an OUD. The objective of the proposed research is to test whether treatment with a GLP-1R agonist can reduce craving in humans with OUD. Understanding how a 'satiety' agent may affect craving and brain responses to drug cues in an OUD population would provide entirely novel information. If liraglutide shows a trend towards efficacy, and safety of the GLP-1R agonist is demonstrated in this population, it would provide an indication to run the second phase, multi-center clinical trial of GLP-1R agonist in OUD patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years
* Diagnosed with an OUD seeking treatment at Caron Treatment Centers (CaronTC) and planning on being enrolled in a residential treatment plan for a minimum of 4 weeks
* Women of childbearing potential must consent to use a medically accepted method of birth control or to abstain from sexual intercourse while in the study
* Able and willing to provide informed consent prior to any study-related activities
* Must be able to read and communicate in English sufficiently to complete all study requirements, including Ecology Momentary Assessment (EMA)

Exclusion Criteria:

* Age < 18 or > 75 years
* Women who are pregnant, planning pregnancy, breastfeeding, or unwilling to use adequate contraceptive measures
* History of angioedema, serious hypersensitivity reaction, or anaphylactic reaction to liraglutide or another glucagon-like peptide-1 receptor (GLP1R) agonist
* Personal or family history of medullary thyroid carcinoma (MTC) or patients with multiple endocrine neoplasia syndrome type 2 (MEN 2) or thyroid nodule
* Type I diabetes or history of diabetic ketoacidosis
* Type II diabetes mellitus
* Hypoglycemia on intake visit (blood glucose < 70 mg/dL)
* End-stage renal failure on dialysis or glomerular filtration rate (GFR) <30 mL/min per 1.73 square meters or previous renal transplant
* Severe hepatic impairment (AST or ALT levels > 3 times upper limit of normal range) or previous liver transplant
* Current or past diagnosis of pancreatitis, gastroparesis, or other severe gastrointestinal disease
* Current or past diagnosis of gallbladder disease or gallstones
* Serious cardiovascular disease within the past 6 months (e.g. uncontrolled hypertension, heart failure, significant cardiac arrhythmias, myocardial infarction, presence of angina pectoris, symptomatic coronary artery disease, deep vein thrombosis, pulmonary embolism, second- or third-degree heart block, mitral valve or aortic stenosis, hypertrophic cardiomyopathy, stroke)
* Severe co-occurring psychiatric disorder (e.g., bipolar disorder, psychotic disorder, schizophrenia) that would, in the opinion of the Principle Investigator or study physician, interfere with participating in the study, such as if the patient needs a higher or different level of care and is going to be transferred out of Caron.
* Suicidal ideation within the past 1 month, or history of suicide attempts within the past 1 year, unless participation is cleared by clinician assessment and/or judgement.
* Treatment with any investigational drug in the one-month preceding the study
* Previous randomization for participation in this trial
* Abnormal physical exam findings, vital signs (blood pressure, heart rate, respiratory rate, body temperature), EKG measurements, and safety lab values that are deemed clinically significant by study physician

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Bunce, PhD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Freet CS, Evans B, Brick TR, Deneke E, Wasserman EJ, Ballard SM, Stankoski DM, Kong L, Raja-Khan N, Nyland JE, Arnold AC, Krishnamurthy VB, Fernandez-Mendoza J, Cleveland HH, Scioli AD, Molchanow A, Messner AE, Ayaz H, Grigson PS, Bunce SC. Ecological momentary assessment and cue-elicited drug craving as primary endpoints: study protocol for a randomized, double-blind, placebo-controlled clinical trial testing the efficacy of a GLP-1 receptor agonist in opioid use disorder. Addict Sci Clin Pract. 2024 Jul 27;19(1):56. doi: 10.1186/s13722-024-00481-7. PMID 39061093

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol was approved for a 3-dose intervention that could continue as a 5-dose intervention; no participants received the latter. All outcomes are reported as the 3-dose intervention.
Pre-assignment Details: Two participants were not randomized due to screening after consent and prior to randomization.
Period: Overall Study
Arm/Group | Investigational Group | Control Group
Started | 12 | 13
Completed | 1 | 8
Not Completed | 11 | 5
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 8 | 3
Not completed — Screen fail after consent | 0 | 1
Not completed — Early withdraw criteria met | 0 | 1
Not completed — Non-compliance/difficulty with staff | 2 | 0

BASELINE CHARACTERISTICS:
Population: Randomized participants in residential treatment for opioid use disorder
Groups:
- Total: Total of all reporting groups
Arm/Group | Investigational Group | Control Group | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.23 (2.04) | 32.03 (2.19) | 33.57 (1.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 11 | 10 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 12 | 24
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 10 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Self-reported Cue-elicited Drug Craving as Measured by Visual Analog Scale (VAS)
Description: Scores are measured on a 0-100 point VAS, where 0= no craving, 100= maximum craving.
Time Frame: Baseline (Day 1), End of the target drug dose (Day 19)
Population: In control group, n=1 did not complete the measure due to technical difficulties. n=7 instead of n=8 reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Investigational Group | Control Group
Number analyzed (Participants) | 1 | 7
score on a scale | -5.00 (NA) — Standard Deviation is not calculable for 1 participant | -13.34 (19.58)

2. Primary Outcome: Change in Ambient Drug Craving Over Time as Measured by Visual Analog Scale (VAS)
Description: Scores are measured on a 0-4 point VAS, where 0= no craving, 4= maximum craving.
Time Frame: Baseline (Day 1), Treatment Days (Days 2-19)
Population: n=1 did not complete entire EMA. n=7 instead of n=8 reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Investigational Group | Control Group
Number analyzed (Participants) | 1 | 7
score on a scale | -0.55 (NA) — Standard Deviation is not calculable for 1 participant | -1.41 (0.99)

3. Secondary Outcome: Change in Blood Pressure
Description: Blood pressure measurements in mmHg. Both systolic and diastolic pressures will be assessed during the study period.
Time Frame: Baseline (Day 1); beginning of each study drug dose (Days 2, 8, 14)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Investigational Group | Control Group
Number analyzed (Participants) | 1 | 8
mmHg
  Systolic Pressure, from Day 2 | 4.00 (NA) — Standard Deviation is not calculable for 1 participant | -0.59 (4.69)
  Systolic Pressure, from Day 8 | 9.00 (NA) — Standard Deviation is not calculable for 1 participant | 2.75 (6.67)
  Systolic Pressure, from Day 14 | 3.75 (NA) — Standard Deviation is not calculable for 1 participant | 2.13 (8.13)
  Diastolic Pressure, from Day 2 | 3.00 (NA) — Standard Deviation is not calculable for 1 participant | 2.56 (6.17)
  Diastolic Pressure, from Day 8 | 2.25 (NA) — Standard Deviation is not calculable for 1 participant | 3.34 (6.61)
  Diastolic Pressure, from Day 14 | 2.75 (NA) — Standard Deviation is not calculable for 1 participant | 4.19 (7.51)

4. Secondary Outcome: Change in Heart Rate
Description: Heart rate measurements in beats per minute.
Time Frame: Baseline (Day 1); beginning of each study drug dose (Days 2, 8, 14)
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Investigational Group | Control Group
Number analyzed (Participants) | 1 | 8
beats per minute
  Day 02 change from baseline | 10.75 (NA) — Standard Deviation is not calculable for 1 participant | -5.78 (5.10)
  Day 08 change from baseline | 20.00 (NA) — Standard Deviation is not calculable for 1 participant | -2.63 (10.98)
  Day 14 change from baseline | 9.75 (NA) — Standard Deviation is not calculable for 1 participant | -3.09 (11.20)

5. Secondary Outcome: Change in Respiratory Rate
Description: Respiratory rate in breaths per minute.
Time Frame: Baseline (Day 1); beginning of each study drug dose (Days 2, 8, 14)
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Investigational Group | Control Group
Number analyzed (Participants) | 1 | 8
breaths per minute
  Day 02 change from baseline | -1.00 (NA) — Standard Deviation is not calculable for 1 participant | 0.08 (2.83)
  Day 08 change from baseline | 0.67 (NA) — Standard Deviation is not calculable for 1 participant | -1.08 (2.74)
  Day 14 change from baseline | 1.33 (NA) — Standard Deviation is not calculable for 1 participant | -0.13 (2.49)

6. Secondary Outcome: Absolute Change in Body Weight
Description: Body weight will be measured in kilograms (kg).
Time Frame: From Day 1 to Day 19
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Investigational Group | Control Group
Number analyzed (Participants) | 1 | 8
kg | 0.27 (NA) — Standard Deviation is not calculable for 1 participant | 1.05 (1.86)

7. Secondary Outcome: Percent Change in Body Weight
Description: Body weight will be measured in kilograms (kg) and change will measured in %.
Time Frame: From Day 1 to Day 19
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Investigational Group | Control Group
Number analyzed (Participants) | 1 | 8
% change | 0.33 (NA) — Standard Deviation is not calculable for 1 participant | 1.38 (2.39)

8. Secondary Outcome: Change in Fasting Blood Samples for Fructosamine
Description: Fructosamine is measured in umol/L
Time Frame: From Day 2 to Day 19
Population: In control group, n=1 could not obtain blood draw for measure. n=7 instead of n=8 reported.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Investigational Group | Control Group
Number analyzed (Participants) | 1 | 7
umol/L | -14.00 (NA) — Standard Deviation is not calculable for 1 participant | 2.71 (21.48)

9. Secondary Outcome: Change in Fasting Blood Samples for HA1c
Description: HA1c is measured in %
Time Frame: From Day 2 to Day 19
Measure: Mean (Standard Deviation); unit: % of total hemoglobin in the blood
Arm/Group | Investigational Group | Control Group
Number analyzed (Participants) | 1 | 8
% of total hemoglobin in the blood | -0.10 (NA) — Standard Deviation is not calculable for 1 participant | 0 (0.11)

10. Secondary Outcome: Frequency of Adverse Events (AE) and Serious Adverse Events (SAE)
Description: Number of participants affected by probable drug-related adverse events.
Time Frame: Days 1-21 and at 30 days post-intervention (Day 49).
Population: Randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Group | Control Group
Number analyzed (Participants) | 12 | 13
Participants
  Participants with drug-related AEs | 5 | 3
  Participants with drug-related SAEs | 1 | 0

11. Other Pre Specified Outcome: Change in Blood Oxygenation Level Response to Visual Opioid Drug Cues in Prefrontal Cortex Using Functional Near Infrared Spectroscopy (fNIRs)
Description: fNIRs indexes regional cerebral oxygenation saturation (%) by optical density (OD). Increased OD indicates increased blood oxygen saturation.
Time Frame: Baseline (Day 1), end of the target drug dose (Day 19)
Population: In placebo group, processing difficulties limited analysis. N=5 reported.
Measure: Mean (Standard Deviation); unit: Optical density (OD)
Arm/Group | Investigational Group | Control Group
Number analyzed (Participants) | 1 | 5
Optical density (OD) | -3.10 (NA) — Standard Deviation is not calculable for 1 participant | -0.58 (0.65)

12. Other Pre Specified Outcome: Rebound Change in Ambient Drug Craving Over Time as Measured by Visual Analog Scale (VAS)
Description: Scores are measured on a 0-4 point VAS, where 0= no craving, 4= maximum craving. Treatment score is the average scores across Days 2-19. Rebound follow up score is the average scores across Days 20-21.
Time Frame: Treatment (averaged across Days 2-19), Rebound follow up (averaged across Days 20-21)
Population: n=1 did not complete entire EMA. n=7 instead of n=8 reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Investigational Group | Control Group
Number analyzed (Participants) | 1 | 7
score on a scale | -0.11 (NA) — Standard Deviation is not calculable for 1 participant | -0.15 (0.47)

13. Other Pre Specified Outcome: Rebound Change in Blood Pressure
Description: Blood pressure measurements in mmHg. Both pressures will be assessed during the study period.
Time Frame: From end of the target drug dose (Day 19) to rebound follow up (Day 21).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Investigational Group | Control Group
Number analyzed (Participants) | 1 | 8
mmHg
  Change in systolic pressure | 11.00 (NA) — Standard Deviation is not calculable for 1 participant | -0.56 (12.45)
  Change in diastolic pressure | 10.25 (NA) — Standard Deviation is not calculable for 1 participant | -1.59 (6.27)

14. Other Pre Specified Outcome: Rebound Change in Heart Rate
Description: Heart rate measurements in beats per minute
Time Frame: From end of the target drug dose (Day 19) to rebound follow up (Day 21).
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Investigational Group | Control Group
Number analyzed (Participants) | 1 | 8
beats per minute | 8.50 (NA) — Standard Deviation is not calculable for 1 participant | -6.31 (8.41)

15. Other Pre Specified Outcome: Rebound Change in Respiratory Rate
Description: Respiratory rate in breaths per minutes.
Time Frame: From end of the target drug dose (Day 19) to rebound follow up (Day 21).
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Investigational Group | Control Group
Number analyzed (Participants) | 1 | 8
breaths per minute | -6.33 (NA) — Standard Deviation is not calculable for 1 participant | -0.67 (2.83)

ADVERSE EVENTS:
Time Frame: 54 days
Description: Subjects were routinely questioned about adverse events and EMR reviewed by nursing and research staff Days 1-21. A follow-up communication was scheduled 30 days (±5 days) after the participant's last treatment day. Participants could be assessed up to 54 days for adverse events.
Arm/Group | Investigational Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 2/12 | 1/13
Other Adverse Events (participants affected / at risk) | 10/12 | 8/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Group (N=12) | Control Group (N=13)
Vasovagal syncope (Vascular disorders) | 1 (1) | 0 (0)
Overdose to illicit drug (General disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Group (N=12) | Control Group (N=13)
Nausea (Gastrointestinal disorders) | 4 (6) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2)
GI/abdominal upset (Gastrointestinal disorders) | 3 (3) | 1 (1)
Decreased appetite (Gastrointestinal disorders) | 1 (2) | 0 (0)
Headache (General disorders) | 3 (4) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (2)
Hiccups (General disorders) | 0 (0) | 1 (1)
Continuing opioid withdrawal (General disorders) | 0 (0) | 1 (1)
Light headed (General disorders) | 1 (1) | 0 (0)
Ringing sensation (General disorders) | 0 (0) | 1 (1)
Knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Discomfort at Dexcom sensor site (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Shakiness, diaphoresis, and tremor (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Night terrors (Psychiatric disorders) | 1 (1) | 0 (0)
Intrusive thoughts or images (Psychiatric disorders) | 1 (1) | 0 (0)
Bleeding under Dexcom sensor (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Bruising at injection site (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin irritation spots (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Insect bite (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-21): https://cdn.clinicaltrials.gov/large-docs/28/NCT04199728/Prot_SAP_000.pdf
  • Informed Consent Form (2024-06-27): https://cdn.clinicaltrials.gov/large-docs/28/NCT04199728/ICF_001.pdf